CLINICAL TRIAL: NCT07404202
Title: Pan HER2: A Multicenter, Non-interventional, Descriptive Study to Assess Assay Concordance of HER2 IHC Testing in Chinese Pan-tumor Patients
Brief Title: A Multicenter, Non-interventional, Descriptive Study to Assess Assay Concordance of HER2 IHC Testing in Chinese Pan-tumor Patients
Acronym: Pan HER2
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673L00020
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pan-tumor(NSCLC, GYN Cancers, BTC and UC)
Keywords: Pan-tumor(NSCLC, GYN cancers, BTC and UC); HER2 assay concordance and interpretation concordance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Retrospectively collect previously archived tissues or slices for HER2 testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NSCLC: Approximately 1,000 non-small cell lung cancer samples are expected to be collected, and 80 patients will be selected to evaluate assay concordance on confusion matrix results between 5 assays and HercepTest.
- BTC: Approximately 500 biliary tract cancer samples are expected to be collected,and 80 patients will be selected to evaluate assay concordance on confusion matrix results between 5 assays and HercepTest.
- GYN: Approximately 450 gynecological cancer samples are expected to be collected, and 80 patients will be selected to evaluate assay concordance on confusion matrix results between 5 assays and HercepTest.
- UC: Approximately 150 urothelial carcinoma samples are expected to be collected,and 80 patients will be selected to evaluate assay concordance on confusion matrix results between 5 assays and HercepTest.

SUMMARY:
This is a multicenter, non-interventional, descriptive study to retrospectively collect solid tumor samples from focused tumor types (NSCLC, GYN cancers, BTC and UC) and assess both assay concordance and interpretation concordance.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional, descriptive study which included about 2100 patients, a mixture of NSCLC, BTC, GYN cancers and UC, from 12 sites with confirmed diagnosis between 2023 Jan and 2025 Sep. This study includes two phases, which are enrollment phase and assessment phase.

In the enrollment phase, all sites will retrospectively collect about 2100 patients (NSCLC ~1,000; BTC ~500; GYN ~450; and UC ~150). Every patient will be tested for HER2 status by 4B5 in local labs. All HER2 results will be reviewed and aligned by a committee of three pathologists using GC algorithms. Based on HER2 results by HercepTest at central lab, patient will be selected for further evaluation in assessment phase.

In assessment phase, a total of 320 patients will be included and selected from enrollment phase to meet sample size requirement which is 80 patients with different HER2 expression level (each 20 cases for IHC 0/1+/2+/3+) in NSCLC, BTC, GYN cancers and UC cohorts.

In Part I Assay performance evaluation, tissue sample of every patient will be sectioned at least 15 slides and send to central labs for assays evaluation. Interpretation results will be reviewed and aligned by a committee of three pathologists using GC algorithms. Assays and performed platform details are listed below: Roche 4B5 in Ventana platform, MXB\Zhongshan\An Biping\Amoy in Ventana (or Leica) platform (5 assays) v.s. HercepTest in Dako platform.

Part II Interpretation concordance evaluation: inter-obsever agreement will be evaluated based on scanned images. Specifically, the first 40 slides (each 10 for 0/1+/2+/3+, each 10 for four disease cohorts) will be selected and digitalized. 36 pathologists, 3 from each site, will be trained for GC interpretation algorithm before joining in the assessment. All slides will be interpreted by all pathologists.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age
2. Male and female patients must have a histological confirmed diagnosis of NSCLC, BTC, GYN cancers, or UC between Jan 01, 2023 and Sep 30, 2025.

   * For GYN cancers, only cervical cancer, endometrial cancer and ovarian cancer should be included. For each gynecological cancer listed above, at least 5 cases need to be enrolled at each expression level (i.e., IHC 0/1+/2+/3+).
3. Patients must have sufficient archived tumor tissue available, with at least 15 slides suitable for HER2 status determination. Both resection or biopsy samples are acceptable. The age limit of archived tissue blocks is 5 years.

Exclusion Criteria:

1. Have a history of other cancers besides NSCLC, BTC, GYN cancers and UC.
2. Specimens of patients that may affect interpretation evaluated by the researcher (e.g., frozen specimens, decalcified specimens, specimens with limited tumor content, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients must have a histological confirmed diagnosis of NSCLC, BTC, GYN cancers, or UC between Jan 01, 2023 and Sep 30, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2026-03-12 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
NPA of HER2 IHC 3+ based on confusion matrix results betwee other assays(Roche 4B5\MXB\Zhongshan\An Biping\Amoy) and HercepTest | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the NPA of HER2 IHC 3+ based on confusion matrix results between other assays(Roche 4B5\MXB\Zhongshan\An Biping\Amoy) and HercepTest
PPA of HER2 IHC 3+ based on confusion matrix results between other assays(Roche 4B5\MXB\Zhongshan\An Biping\Amoy) and HercepTest | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the PPA of HER2 IHC 3+ based on confusion matrix results between other assays (Roche 4B5\MXB\Zhongshan\An Biping\Amoy) and HercepTest

SECONDARY OUTCOMES:
Inter-observer concordance in binary HER2 negative (IHC 0/1+/2+) and positive status (IHC3+); | From first slides interpreted to Interpretation concordance evaluation end，up to approximately 6 month
  To assess the Inter-observer concordance in binary HER2 negative (IHC 0/1+/2+) and positive status (IHC3+);
Inter-observer concordance in binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+); | From first slides interpreted to Interpretation concordance evaluation end，up to approximately 6 month
  To assess the Inter-observer concordance in binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+);
Inter-observer concordance in four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0 | From first slides interpreted to Interpretation concordance evaluation end，up to approximately 6 month
  To assess the Inter-observer concordance in four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0
OPA of HER2 IHC 3+ based on confusion matrix results between other assays and HercepTest | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the OPA of HER2 IHC 3+ based on confusion matrix results between other assays and HercepTest
Cohen's kappa of HER2 IHC 3+ based on confusion matrix results between other assays and HercepTest | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the Cohen's kappa of HER2 IHC 3+ based on confusion matrix results between other assays and HercepTest
NPA of binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+), and four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0 based on confusion matrix results between other assay and HercepTest, overall and by disease cohort | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the NPA of binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+), and four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0 based on confusion matrix results between other assay and HercepTest, overall and by disease cohort
PPA of binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+), and four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0 based on confusion matrix results between other assay and HercepTest, overall and by disease cohort | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the PPA of binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+), and four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0 based on confusion matrix results between other assay and HercepTest, overall and by disease cohort
OPA of binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+), and four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0 based on confusion matrix results between other assay and HercepTest, overall and by disease cohort | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the OPA of binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+), and four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0 based on confusion matrix results between other assay and HercepTest, overall and by disease cohort
Cohen's kappa of binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+), and four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0 based on confusion matrix results between other assay and HercepTest, overall and by disease cohort | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the Cohen's kappa of binary HER2 (IHC 0/1+) v.s. HER2 (IHC 2+/3+), and four category HER2 IHC 3+ vs. IHC 2+ vs. IHC 1+ vs. IHC 0 based on confusion matrix results between other assay and HercepTest, overall and by disease cohort
NPA of HER2 IHC 2+/3+ (IHC 1+ in GYN cancers) based on confusion matrix results between other assay and HercepTest, overall and by disease cohort | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the NPA of HER2 IHC 2+/3+ (IHC 1+ in GYN cancers) based on confusion matrix results between other assay and HercepTest, overall and by disease cohort
PPA of HER2 IHC 2+/3+ (IHC 1+ in GYN cancers) based on confusion matrix results between other assay and HercepTest, overall and by disease cohort | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the PPA of HER2 IHC 2+/3+ (IHC 1+ in GYN cancers) based on confusion matrix results between other assay and HercepTest, overall and by disease cohort
OPA of HER2 IHC 2+/3+ (IHC 1+ in GYN cancers) based on confusion matrix results between other assay and HercepTest, overall and by disease cohort | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the OPA of HER2 IHC 2+/3+ (IHC 1+ in GYN cancers) based on confusion matrix results between other assay and HercepTest, overall and by disease cohort
Cohen's kappa of HER2 IHC 2+/3+ (IHC 1+ in GYN cancers) based on confusion matrix results between other assay and HercepTest, overall and by disease cohort | From the assessment phase start to the final slides interpreted，up to approximately 6 month
  To assess the Cohen's kappa of HER2 IHC 2+/3+ (IHC 1+ in GYN cancers) based on confusion matrix results between other assay and HercepTest, overall and by disease cohort

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient- level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes,indicates that AZ are accepting requests for IPD,but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitment at made to the EFPIA Pharma Data Sharing Principles .For details of our timeline please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment vivli.org. Signed Data Usage Agreement(non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/